CLINICAL TRIAL: NCT02189330
Title: A Phase 1, Open-Label, Randomized, 2-Cohort, Crossover, Single Dose Study to Estimate the Relative Bioavailability of PF 06291826 (Tafamidis) Following Administration of Two Oral Formulations Versus Commercial Capsule in Healthy Subjects Under Fasted Conditions
Brief Title: A Study To Estimate How Much Tafamidis Created In Different Ways Can Be Measured in Blood Samples
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461030
Record Dates: First submitted 2014-05-15; First posted 2014-07-14 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Tafamidis (Experimental)
  Interventions: Drug: Tafamidis
- Tafamudus Free Acid (Experimental)
  Interventions: Drug: Tafamidis
- 20 mg new soft gelatin capsule (Experimental)
  Interventions: Drug: Tafamidis
- 4 capsules of 20 mg tafamidis of commercial formulation (Experimental)
  Interventions: Drug: Tafamidis
- 4 capsules of 12.2 mg tafamidis of free acid tablet (Experimental)
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — 20 mg of current commercial formulation.
  Arms: Tafamidis
Drug: Tafamidis — 12.2 mgA free acid tablet.
  Arms: Tafamudus Free Acid
Drug: Tafamidis — 20 mg new soft gelatin capsule.
  Arms: 20 mg new soft gelatin capsule
Drug: Tafamidis — 4 capsules of 20 mg tafamidis of current commercial formulation.
  Arms: 4 capsules of 20 mg tafamidis of commercial formulation
Drug: Tafamidis — 4 capsules of 12.2 mg tafamidis of free acid tablet..
  Arms: 4 capsules of 12.2 mg tafamidis of free acid tablet

SUMMARY:
All subjects in this study will be given tafamidis. After swallowing a single pill of tafamidis, measurements including blood samples will be compared to see if tafamidis made in different ways is about the same. After approximately 28 days subjects will be given another pill of tafamidis and the study measurements will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-child bearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 and total body weight more than 50 kg (110 lbs).

Exclusion Criteria:

* Blood pressure at screening visit of greater than 140 mm Hg (systolic) or 90 mg Hg (diastolic).
* Use of prescription or nonprescription drugs supplements within 7 days prior to 7 days of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 168 hours
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 168 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 168 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461030&StudyName=A%20Study%20To%20Estimate%20How%20Much%20Tafamidis%20Created%20In%20Different%20Ways%20Can%20Be%20Measured%20in%20Blood%20Samples